CLINICAL TRIAL: NCT00488995
Title: A Phase 2 Study To Evaluate The Safety, Tolerability, Virologic And Immunologic Effect Of Single-Dose CP-675,206 In Patients Infected With Human Immunodeficiency Virus
Brief Title: Safety And Efficacy Study Of CP-675,206 In HIV-Infected Patients
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: A3671029
Record Dates: First submitted 2007-06-19; First posted 2007-06-20 (Estimated); Last update posted 2015-03-11 (Estimated); Status verified 2015-03

CONDITIONS: Human Immunodeficiency Virus
Keywords: HIV Therapeutic Vaccine
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — tremelimumab

INTERVENTIONS:
Drug: CP-675,206

SUMMARY:
The purpose of this study is to determine if CP-675,206, a monoclonal antibody to CTLA4, is safe and well-tolerated, reduces viral load, and improves immune function in patients infected with HIV.

ELIGIBILITY:
Inclusion Criteria:

* HIV infected man or woman at least 18 years of age who is available for a follow up period of at least 3 months
* Has been on a stable antiretroviral regimen for ≥3 months and willing to remain on current antiretroviral regimen for an additional 3 months or has been off of antiretroviral therapy for at least 8 weeks and willing to remain off of antiretroviral therapy for another 3 months
* Plasma HIV 1 RNA ≥5,000 copies/mL measured by Roche Amplicor HIV 1 Monitor at the screening visit
* CD4 T-cells ≥200 cells/mm3

Exclusion Criteria:

* History of, or significant evidence of risk for, chronic inflammatory or autoimmunedisease (eg, Addison's disease, asthma, celiac disease, multiple sclerosis, Graves disease, Hashimoto's thyroiditis, inflammatory bowel disease, psoriasis, rheumatoid arthritis, systemic lupus erythematosus, etc)
* History of inflammatory bowel disease (eg, Crohn's disease or ulcerative colitis), celiac disease, or other chronic gastrointestinal conditions associated with diarrhea, or current acute colitis of any origin, and any history of diverticulitis (even a single episode) or evidence of diverticulitis at baseline, including evidence limited to CT-scan only
* Exposure within the previous 3 months to a drug known to have immunomodulatory effects (eg, IL 2)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-07

PRIMARY OUTCOMES:
Maximum reduction in HIV plasma RNA between Baseline and Week 12 Maximum increase in CD4+ cell count between Baseline and Week 12

SECONDARY OUTCOMES:
Change from baseline in CD8+ cell count, CD4/CD8, and lymphocyte phenotype through Week 12

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3671029&StudyName=Safety+And+Efficacy+Study+Of+CP%2D675%2C206+In+HIV%2DInfected+Patients